CLINICAL TRIAL: NCT02538601
Title: Enhanced Smoking Cessation Intervention for Smokers Exposed to the WTC Disaster
Brief Title: Enhanced Smoking Cessation Intervention for Smokers Exposed to the World Trade Center (WTC) Disaster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-1605
Record Dates: First submitted 2015-08-12; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Cigarette Smoking; Post Traumatic Stress Disorder; Signs and Symptoms, Respiratory
Keywords: Post Traumatic Stress Disorder; PTSD; Cigarette Smoking; Lower Respiratory Symptoms; Cognitive Behavioral Therapy; CBT; Transdiagnostic Treatments; World Trade Center
MeSH Terms: conditions — Cigarette Smoking; Stress Disorders, Post-Traumatic; Signs and Symptoms, Respiratory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-A (Experimental): An 8-session, CBT-based group smoking cessation program (CBT-A) enhanced with transdiagnostic skills for the management of anxiety and fear-based avoidance behaviors.
  Interventions: Behavioral: CBT-A
- CBT-S (Active Comparator): An 8-session, CBT-based, traditional group CBT based smoking cessation program.
  Interventions: Behavioral: CBT-S

INTERVENTIONS:
Behavioral: CBT-A — CBT-A was an 8-session (1.5 hours/session) group treatment for quitting smoking comprised of an optimized protocol that incorporated all elements of the CBT-S treatment plus skills for reducing PTSD/anxiety symptoms and improving tolerance to withdrawal. The CBT-A intervention included skills based on a transdiagnostic approach: (1) repeated interoceptive exposures to feared bodily sensations (e.g., dizziness, racing heart); (2) corrective information about anxiety and cognitive restructuring of catastrophic misinterpretations of somatic sensations (e.g., "I will lose control."); and (3) use of graduated in-vivo exposure to feared and avoided situational experiences related to anxiety, WTC-related PTSD triggers, and smoking (e.g., going to lower Manhattan; driving without smoking).
  Arms: CBT-A
Behavioral: CBT-S — CBT-S was an adapted group-based CBT smoking cessation treatment delivered in 8 sessions (1.5 hours/session) based on the most recent clinical practice guidelines from the United States Department of Health and Human Services (USDHHS), Treating Tobacco Use and Dependence. Standard cessation elements included psychoeducation on reasons for smoking and barriers to quitting, enlisting social support, monitoring and tapering cigarette use, and counseling regarding high-risk smoking situations and unhelpful ways of thinking about smoking and abstinence. The treatment was similar to protocols used in other smoking cessation research.
  Arms: CBT-S

SUMMARY:
The purpose of this study was to test the efficacy of a CBT-based smoking cessation treatment enhanced with transdiagnostic skills for the management of anxiety and fear-based avoidance behaviors (CBT-A) relative to a standard CBT-based smoking cessation treatment (CBT-S) for smokers with elevated PTSD symptoms who were exposed to the 9/11 World Trade Center disaster. The investigators hypothesized that the CBT-A treatment would yield more favorable outcomes with regard to smoking abstinence as well as improvements in PTSD and respiratory symptoms over a 6-month follow-up period.

DETAILED DESCRIPTION:
Respiratory illness and post-traumatic stress disorder (PTSD) are the primary health sequelae of the World Trade Center (WTC) disaster on September 11th 2001 and are often comorbid. Cigarette smoking is a modifiable health behavior associated with both lower respiratory symptoms (LRS) and PTSD. Smoking cessation programs are considered the crucial front-line intervention for smokers with pulmonary problems. Unfortunately, trauma exposed smokers with elevated PTSD symptoms have greater difficulty quitting, are more likely to fail standard cessation programs, and are more likely to relapse than smokers with other anxiety disorders and those without mental illness. Interventions that concurrently target mechanisms thought to maintain the comorbidity between PTSD and LRS (e.g., anxious reactivity to nicotine withdrawal, smoking to reduce negative affect) may offer a means of improving smoking quit rates in trauma exposed populations. Thus, the purpose of this study was to test the efficacy of a combined CBT smoking cessation treatment enhanced with transdiagnostic skills for the management of anxiety and fear-based avoidance behaviors (CBT-A). The investigators randomized 90 WTC disaster exposed daily smokers with elevated PTSD symptoms to either CBT-A (N=44) or a standard CBT-based smoking cessation program (CBT-S; N=46). Participants were followed up to six months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* smoking at least five cigarettes per day
* reporting interest in smoking cessation treatment
* direct exposure to the WTC disaster (e.g., responding to the event or witnessing the event in person)
* scoring >30 on the Posttraumatic Stress Disorder Checklist

Exclusion Criteria:

* current participation in another smoking cessation treatment
* alcohol dependence within the last six months
* serious mental illness (e.g., psychosis, mania)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Session 8 7-day point prevalence cigarette abstinence | Session 8: on average 2 weeks post-quit day
  A dichotomized outcome (yes/no) configured based on biochemically verified 7 day smoking abstinence via Saliva cotinine (cutoff value of 10 ng/ml) and carbon monoxide (CO) analysis of breath samples with a Vitalograph Breathco CO monitor.
6-month Follow-up 7-day point prevalence cigarette abstinence | 6-month follow-up
  A dichotomized outcome (yes/no) configured based on biochemically verified 7 day smoking abstinence via Saliva cotinine (cutoff value of 10 ng/ml) and carbon monoxide (CO) analysis of breath samples with a Vitalograph Breathco CO monitor.

SECONDARY OUTCOMES:
Change in WTC related post-traumatic stress disorder (PTSD) symptoms | Baseline and 2-weeks post-quit attempt
  Assessed via self-report (PTSD Checklist Specific Stressor; PCL-S)
6-month change in WTC related post-traumatic stress disorder (PTSD) symptoms | Baseline and 6-month follow-up
  Assessed via self-report (PTSD Checklist Specific Stressor; PCL-S)
Change in lower respiratory symptoms | Baseline and 2-weeks post-quit attempt
  Assessed via self-report
6-month change in lower respiratory symptoms | Baseline and 6-month follow-up
  Assessed via self-report
Change in average daily cigarettes smoked | Baseline and 2-weeks post-quit attempt
  Average number of cigarettes smoke per day in the past 7 days assessed via Time Line Follow-Back (TLFB) for Daily Cigarette Use
6-month change in average daily cigarettes smoked | Baseline and 6-month follow-up
  Average number of cigarettes smoke per day in the past 7 days assessed via Time Line Follow-Back (TLFB) for Daily Cigarette Use

CONTACTS AND LOCATIONS:
Overall Officials: Roman Kotov, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Putnam Hall, Stony Brook, New York, United States

REFERENCES:
- [Derived] Waszczuk MA, Li X, Bromet EJ, Gonzalez A, Zvolensky MJ, Ruggero C, Luft BJ, Kotov R. Pathway from PTSD to respiratory health: Longitudinal evidence from a psychosocial intervention. Health Psychol. 2017 May;36(5):429-437. doi: 10.1037/hea0000472. Epub 2017 Mar 9. PMID 28277702